CLINICAL TRIAL: NCT02251262
Title: Assessment of Diagnostic Accuracy of 18FDG-PET-CT in Patients With Suspicion of Pacing or Defibrillation Lead Infection: a Prospective Multi-center Study
Brief Title: Diagnostic Accuracy of 18FDG-PET-CT for Pacing or Defibrillation Lead Infection
Acronym: ENDOTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUBX 2013/31
Record Dates: First submitted 2014-09-24; First posted 2014-09-29 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Infections of the Implanted Material; Endocarditis
Keywords: Pacemaker; Endocarditis; 18FDG-PET-CT; Diagnostic accuracy; Pacing or defibrillation lead
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whole-body 18FDG-PET-CT scan (Experimental): 18FDG-PET-CT exam will be performed in patients, with suspicion of pacing or defibrillation lead infection, hospitalized in cardiology unit.
  Interventions: Device: Whole-body 18FDG-PET-CT scan

INTERVENTIONS:
Device: Whole-body 18FDG-PET-CT scan — 18FDG-PET-CT exam will be performed in patients, with suspicion of pacing or defibrillation lead infection, hospitalized in cardiology unit.

SUMMARY:
With aging of the general population and broadening indications, the number of pacemaker recipients is steadily increasing. The incidence of infections of the implanted material, a dreaded major complication, is also rising. The diagnosis is evident in presence of an abscessed pocket, cutaneous breakthrough of the pulse generator or vegetations attached to the lead. On the other hand, a proportion of patients present with less specific clinical manifestations and a pacemaker recipient may be recurrently hospitalized for an infectious disorder of unknown origin despite detailed investigations. Without proof of lead infection, removal of the system without confirmation of its infection is usually proposed, despite the known morbidity and mortality associated with the extraction procedure (0.5 to 2%). Positive culture of the leads implies that the leads were involved in the infectious process. In recent years, 18FDG-PET-CT scan has made promising contributions in different areas including imaging to detect infection at different organ sites. Absence of hyperfixation of the lead, identified by 18FDG-PET/CT scan may be an accurate sign of absence of pacing system infection.

The extraction of intracardiac implanted material, when it is indicated by the current standard strategy, may result in negative bacteriological cultures in 10 to 25% of patients, even when they did not receive antibiotics before extraction.

The hypothesis of the study is that a new strategy adding 18FDG-PET-CT to the current strategy may avoid or reduce these false-positives.

Therefore it is hypothesized that the sensitivity of 18FDG-PET-CT will be high enough to avoid unnecessary extractions of uninfected leads, resulting in a high negative predictive value of the new diagnostic strategy incorporating 18FDG-PET-CT. The present study aims at providing valid estimates of diagnostic accuracy parameters of 18FDG-PET-CT, especially its sensitivity.

For this clinical study, firstly, 18FDG-PET-CT exam will be performed in patients, with suspicion of pacing or defibrillation lead infection, hospitalized in cardiology unit; secondarily, an intervention for the extraction of the intra-cardiac material, under general anesthesia, will be practiced and then a bacteriological culture for extracted material will be required.

The end of study visit is complete the last day of material extraction. The follow up will last 2 to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age > 18 years
* Patient referred for extraction of cardiac material (box and lead(s)) in the context of suspicion of material infection, including a patient with pocket infection.
* Possibility of carrying out PET-CT no more than 48 hours before extraction (or, exceptionally, no more than 7 days if the patient is not under antibiotic therapy).
* Informed written consent
* Affiliation to a social security system

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with recent implantation (less than 2 months)
* Subjects placed under judicial protection
* Subjects participating in another study that includes an exclusion period on-going at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
A semi-quantitative visual interpretation of 18FDG-PET-CT in the diagnosis of infection of intracardiac device. | up to 48 hours after inclusion (exceptionally, up to 7 days if the patient is not under antibiotic therapy)
  Index tests will be interpreted by nuclear medicine physician from the center where the patient was included with a semi-quantitative visual score.
  Moreover, all 18FDG-PET-CT recordings will be sent to the coordinating center for centralized interpretation blind to the preceding one.
  All 18FDG-PET-CT recordings will be stored until interpretation, and not used for the clinical management of the patient.
  Index test interpretations will be carried out blind to any other information on the patient (clinical, biology,…).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BORDACHAR, MD, Principal Investigator — University Hospital, Bordeaux; Paul PEREZ, MD, PhD, Study Chair — University Hospital, Bordeaux
Locations (6):
- France (6):
  - CHU de Grenoble - Hôpital A. Michallon, Grenoble
  - CHRU de Lille - Hôpital R. Salengro, Lille
  - AP-HM - Hôpital La Timone, Marseille
  - CHU de Bordeaux, Pessac
  - Clinique Pasteur, Toulouse
  - CHU de Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy